CLINICAL TRIAL: NCT03037398
Title: Closed Loop Programming Evaluation Using External Responses for Deep Brain Stimulation
Acronym: CLOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A4063
Record Dates: First submitted 2017-01-12; First posted 2017-01-31 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel Arm (Active Comparator): Programming completed by a novel method
  Interventions: Device: Vercise Deep Brain Stimulation System
- Standard of Care Arm (Other): Programming completed as Standard of care
  Interventions: Device: Vercise Deep Brain Stimulation System

INTERVENTIONS:
Device: Vercise Deep Brain Stimulation System

SUMMARY:
The objective of this study is to evaluate the performance of novel DBS programming methods compared to traditional programming methods.

ELIGIBILITY:
Key Inclusion Criteria:

* Implanted bilaterally in STN or GPi with a Vercise™ DBS system for Parkinson's disease, including directional leads, for at least four months and programming optimized according to standard of care with no changes to electrode configuration of primary settings for at least four weeks.
* Able to understand the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
* Be at least 18 years of age.
* Device must have been implanted on label or must be on label by the time the subject gets enrolled.

Key Exclusion Criteria:

* Any significant psychiatric problems, including unrelated clinically significant depression as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Difference in time to program between the two arms at Programming Visit | at least four months post implant

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (3):
- Germany (3):
  - University Berlin, Charite Virchow Standort, Wedding, Berlin
  - Universitaetsklinik Eppendorf, Hamburg
  - Universitätsklinikum Campus Kiel, Kiel

IPD SHARING:
Plan to Share IPD: No